CLINICAL TRIAL: NCT02795624
Title: Vascular Aging in Flight Attendants With Occupational Secondhand Smoke Exposure
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Other Study IDs: Pro00042101
Record Dates: First submitted 2016-01-27; First posted 2016-06-10 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Vascular Aging; Secondhand Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Flight attendants: Flight attendants
  Interventions: Procedure: Spirometry; Procedure: Pulse Wave Analysis; Procedure: Peripheral arterial tonometry

INTERVENTIONS:
Procedure: Spirometry — Test is done to assess how well the lungs work by measuring how much air is inhaled, how much is exhaled, and how quickly it is exhaled.
  Other Names: Breathing test
Procedure: Pulse Wave Analysis — It is a non-invasive assessment of the pulse character
  Other Names: PWA; Arterial stiffness test
Procedure: Peripheral arterial tonometry — It is a non-invasive method to measure endothelial dysfunction.
  Other Names: Endothelial function test

SUMMARY:
Specific Aim 1. Characterize the long-term effects of secondhand smoke (SHS) on vascular health in pre-ban flight attendants (FAs). Investigators will measure arterial stiffness (pulse wave velocity and augmentation index) and endothelial dysfunction (reactive hyperemia index) in the pre-ban FA cases, and compare to the cardiovascular risk-factor matched Framingham controls.

It is hypothesized that pre-ban FA cases have increased arterial stiffness (higher pulse wave velocity and higher augmentation index) and increased endothelial dysfunction (lower reactive hyperemia index) compared to Framingham controls.

Specific Aim 2. Determine the extent in which remote pre-ban SHS exposure (hours) is associated with increased arterial stiffness or endothelial dysfunction.

Investigators hypothesize that pre-ban SHS exposure is positively associated with both increased arterial stiffness and increased endothelial dysfunction.

Specific Aim 3. Investigators will calculate the cardiovascular risk scores (Framingham, Reynolds, and ASCVD) by using subjects' age, blood pressure, family history, lipid panel, and highly sensitive C-reactive protein. Investigators will explore the association of the risk scores with measures of vascular aging (arterial stiffness and endothelial dysfunction). These scores do not include SHS exposure. Investigators will also test the additive value of SHS exposure in increasing arterial stiffness and endothelial dysfunction using the risk scores as an adjustment value.

It is hypothesized that the cardiovascular risk scores are associated with vascular aging (arterial stiffness and endothelial dysfunction), and that the association between SHS exposure and vascular aging remains significant after adjusting for the cardiovascular risk scores.

The significance of this proposal and impact will be (1) mechanistic insights into how remote SHS exposure leads to hypertension and vascular stiffness, (2) increased understanding of how SHS exposure can increase risk of cardiovascular disease, which is the number one cause of death in the United States.

DETAILED DESCRIPTION:
The investigators propose a cohort study, in which investigators will assess for evidence of accelerated vascular aging in 300 pre-ban FAs with pre-ban SHS exposure, and compare their vascular measures of arterial stiffness and endothelial dysfunction to those of age and risk-factor matched Framingham controls. It is hypothesized that pre-ban FAs have increased arterial stiffness and endothelial dysfunction compared to the Framingham subjects, related to SHS exposure.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age and older;
* Flight attendant, including current or past employment with the airlines;
* Non-smoking flight attendant (current and prior, defined as smoking <100 cigarettes in your lifetime);
* Exposed to secondhand tobacco smoke for at least one year, while working on the aircrafts

Exclusion Criteria:

* History of Raynaud's syndrome
* Had mastectomy or arm/hand abnormality in which blood pressure cannot be measured on the arm

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Flight attendants that are 40 years of age and older, with prior occupation secondhand smoke (SHS) exposure pre- and post- smoking ban.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-02; Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Endothelial Dysfunction (RHI) | Baseline
  Reactive hyperemia index (RHI) will be measured by Peripheral Arterial Tonometry, which reflects endothelial dysfunction
Arterial Stiffness (PWV) | Baseline
  During Pulse Wave analysis, pulse wave velocity (PWV) will be measured
Arterial Stiffness (AIx) | Baseline
  During Pulse Wave analysis, augmentation index (AIx) wil be measured

SECONDARY OUTCOMES:
Cardiovascular risk | Baseline
  Framingham 10-year risk
Cardiovascular risk | Baseline
  Reynolds 10-year risk
Cardiovascular risk | Baseline
  American Heart Association/ACC 10-year risk
Cardiovascular risk | Baseline
  American Heart Association/ACC Lifetime risk

CONTACTS AND LOCATIONS:
Overall Officials: C.Noel Bairey Merz, MD, FACC, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Women's Heart Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes